CLINICAL TRIAL: NCT01212549
Title: Open Label, Randomized Comparison of Two Schemes of Cryosurgery and Imiquimod Combination Treatment for Basal Cell Carcinoma of the Skin
Brief Title: Comparison of Two Schemes of Cryosurgery and Imiquimod Combination Treatment for Basal Cell Carcinoma
Acronym: IMCXvsCIMT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Ioannis Bassukas, Associate Professor of Dermatology, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 524270910
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma; cryosurgery; imiquimod; immunocryosurgery
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunocryosurgery (Active Comparator): 2 weeks imiquimod, cryosurgery (open spray liquid nitrogen, 2 cycles, 15 secs each), 3 weeks imiquimod
  Interventions: Procedure: Immunocryosurgery
- Cryoimmunotherapy (Active Comparator): Cryosurgery (open spray liquid nitrogen, 2 cycles, 15 secs each), 5 weeks imiquimod
  Interventions: Procedure: Cryoimmunotherapy

INTERVENTIONS:
Procedure: Immunocryosurgery — 2 weeks imiquimod, cryosurgery (open spray liquid nitrogen, 2 cycles, 15 secs each), 3 more weeks imiquimod
  Arms: Immunocryosurgery
Procedure: Cryoimmunotherapy — Cryosurgery(open spray liquid nitrogen, 2 cycles, 15 secs each), followed by 5 weeks imiquimod
  Arms: Cryoimmunotherapy

SUMMARY:
To compare the effectiveness of two application schemes of cryosurgery during a 5 week course of topical imiquimod i.e. cryosurgery at the end of the second week of imiquimod followed by 3 more weeks of imiquimod (immunocryosurgery) versus cryosurgery at day 0 followed by 5 weeks of topical imiquimod (cryoimmunotherapy)

DETAILED DESCRIPTION:
Comparison of efficacy

* Number of patients: N=40
* Arms: Two equal arms (20 patients each)
* Inclusion criteria: Basal cell carcinoma of the skin proven with biopsy
* Exclusion criteria: (1) Size of the tumors >5cm; (2) Distance from the eyelid <0,5cm; (3)Number of tumors >5
* Interim analysis: When at least 10 patients are included in each arm or at the end of the first year of the study

The patients will be randomized in 2 groups Group 1 (Immunocryosurgery) and Group 2 (Cryoimmunotherapy)

Treatment protocols:

Group 1 (Immunocryosurgery): Patients will apply imiquimod daily for 14 days on the tumor and a rim of 2mm around the tumor. On day 14 a session of mild cryosurgery (2 cycles of 15 seconds, with open spray liquid nitrogen) will be applied and the patients will continue application of imiquimod for another 3 weeks before being evaluated again.

Group 2 (Cryoimmunotherapy): Patients will be submitted into cryosurgery (2 cycles of 15 seconds, with open spray liquid nitrogen) and subsequently will apply imiquimod on the tumor and a rim of 2mm around the tumor for 5 weeks in total. They will be evaluated in week 2 and 5.

Patients from both groups will be evaluated at 1, 3, 6, 12 months after termination of imiquimod treatment. In case of clinical relapse, it will be confirmed by biopsy and all the patients will treated with immunocrysurgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven basal cell carcinoma of the skin
* Size <5cm
* Number of tumors <5 cm
* Distance from eyelids, mouth 0,5cm

Exclusion Criteria:

* Size >5cm
* Number of tumors > or =5
* Distance from eyelids or mouth < or =0.5cm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of immunocryosurgery and cryoimmunotherapy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis D Bassukas, Professor, Principal Investigator — Medical School, University of Ioannina
Locations (1):
- Department for Skin and Venereal Diseases, University Hospital, Ioannina, Greece

REFERENCES:
- [Background] Gaitanis G, Nomikos K, Vava E, Alexopoulos EC, Bassukas ID. Immunocryosurgery for basal cell carcinoma: results of a pilot, prospective, open-label study of cryosurgery during continued imiquimod application. J Eur Acad Dermatol Venereol. 2009 Dec;23(12):1427-31. doi: 10.1111/j.1468-3083.2009.03224.x. Epub 2009 Jun 25. PMID 19555364
- [Background] Bassukas ID, Gaitanis G. Combination of cryosurgery and topical imiquimod: does timing matter for successful immunocryosurgery? Cryobiology. 2009 Aug;59(1):116-7. doi: 10.1016/j.cryobiol.2009.04.011. Epub 2009 May 6. No abstract available. PMID 19426725
- [Background] Bassukas ID, Gamvroulia C, Zioga A, Nomikos K, Fotika C. Cryosurgery during topical imiquimod: a successful combination modality for lentigo maligna. Int J Dermatol. 2008 May;47(5):519-21. doi: 10.1111/j.1365-4632.2008.03562.x. PMID 18412875
- [Background] Gaitanis G, Mitsou G, Tsiouri G, Alexis I, Bassukas ID. Cryosurgery during imiquimod cream treatment ("immunocryosurgery") for Bowen's disease of the skin: a case series. Acta Derm Venereol. 2010 Sep;90(5):533-4. doi: 10.2340/00015555-0896. No abstract available. PMID 20814639